CLINICAL TRIAL: NCT00431158
Title: ARDSnet Protocol vs. the Open Lung Approach for the Ventilatory Management of Severe, Established ARDS: A Global Randomized Controlled Trial
Brief Title: ARDSnet Protocol vs. Open Lung Approach in ARDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Robert M. Kacmarek, Professor of Anesthesia, Director of Respiratory Care Services, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-P-001878; BWH IRB Assurance #FWA00000484
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Acute Respiratory Distress Syndrome; ARDS; Respiratory failure; Mechanical Ventilation; Positive end expiratory pressure; Lung recruitment maneuver
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): ARDSnet Protocol
  Interventions: Other: Different Mechanical Ventilation Protocols
- 2 (Active Comparator): OLA Protocol
  Interventions: Other: Different Mechanical Ventilation Protocols

INTERVENTIONS:
Other: Different Mechanical Ventilation Protocols — OLA Group: Open lung approach protocol and recruitment maneuvers
  ARDSnet Group: ARDSnet protocol

SUMMARY:
Many patients with Acute Respiratory Distress Syndrome or ARDS need breathing support that is provided by a machine called a ventilator or respirator. The purpose of this study is to find out if a new method of setting the ventilator for patients with severe ARDS is better than the standard, commonly used way of setting the ventilator.

DETAILED DESCRIPTION:
The ARDSnet protocol is the current, standard of care for ARDS. Mechanical ventilation is managed using low tidal volumes, relatively high respiratory rates, with oxygenation managed according to PEEP and FIO2 relationships as defined in a table. This study compares the ARDSnet protocol with an open lung approach to mechanical ventilation. The open lung approach uses a technique to recruit collapsed lung areas and then uses the lowest PEEP level that prevents recollapse of recruited lung units. The best PEEP level is determined by a decremental PEEP trial involving a series of pressure measurements taken after the recruitment maneuver. Both the ARDSnet protocol and the open lung approach require low tidal volumes and plateau pressures.

Evidence suggests that using a mechanical ventilation strategy of recruitment maneuvers (to open the collapsed lung) followed by high PEEP (to prevent collapse of the opened lung) with control of transpulmonary pressure through lower plateau pressures would maximize homogeneity within the lung and as such, minimize shearing forces in the lung parenchyma, thus improving ventilation and outcome in mechanically ventilated ARDS patients.

ELIGIBILITY:
Inclusion Criteria:

* Intubated and mechanically ventilated
* Diagnosis of ARDS using American-European consensus criteria
* Enrollment in study < 48 hours since diagnosis of ARDS
* For 12-36 hrs. (ideally 12-24 hrs) after diagnosis of ARDS, patient must be ventilated as follows: Volume A/C, Tidal volume of 4-8 ml/kg PBW, Plateau pressure ≤ 30 cmH2O, PEEP/FIO2 adjustments using ARDSnet table, Ventilator rate to keep PaCO2 = 35-60 mmHg
* During the 12-36 hour(ideally 12-24 hr) period, PaO2/FIO2 must remain < 200 mm Hg for an ABG obtained 30 minutes after placement on the following specific ventilator settings: Volume A/C, Tidal volume = 6 ml/kg PBW, Plateau pressure ≤ 30 cmH2O, Inspiratory time ≤ 1 second, PEEP ≥ 10 cmH2O, FIO2 ≥ 0.5, Ventilator rate to keep PaCO2 = 35-60 mmHg
* No lung recruitment maneuvers or adjunct therapy.
* Total time on mechanical ventilation < 96 hrs. at time of randomization.

Exclusion Criteria:

* Age < 18 years or > 80 years
* Weight < 35 kg PBW
* Body mass index > 60
* Intubated 2° to acute exacerbation of a chronic pulmonary disease
* Acute brain injury (ICP > 18 mmHg)
* Immunosuppression 2° to chemo- or radiation therapy
* Severe cardiac disease(one of the following): New York Heart Association Class 3 or 4, acute coronary syndrome or persistent ventricular tachyarrhythmias
* Positive laboratory pregnancy test
* Sickle cell disease
* Neuromuscular disease
* High risk of mortality within 3 months from cause other than ARDS, e.g. cancer
* More than 2 organ failures (not including pulmonary system)
* Documented lung barotrauma, i.e. chest tube placement other than for fluid drainage
* Persistent hemodynamic instability or intractable shock
* Penetrating chest trauma
* Enrollment in another interventional study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2007-01; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
60 day mortality | 60 days

SECONDARY OUTCOMES:
ICU mortality | Duration of ICU stay
Hospital mortality | Duration of hospital stay
28 day mortality | 28 days
180 day mortality | 180 days
365 day mortality | 365 days
Ventilator free days | Hospital stay
Length of ICU stay | Duration of ICU stay
Development of extra-pulmonary organ failures | Duration of hospital stay
Duration of hospitalization | Duration of hospital stay
Incidence of barotrauma | Duration of hospital stay
Systemic inflammatory mediator levels | Duration of hospital stay
Lung function 6 months after discharge | 6 months
Lung function 12 months after discharge | 12 months
Need for rescue therapy | Duration of hospital stay
Ventilation associated pneumonia rate | Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Kacmarek, Ph.D., R.R.T, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kacmarek RM, Villar J, Sulemanji D, Montiel R, Ferrando C, Blanco J, Koh Y, Soler JA, Martinez D, Hernandez M, Tucci M, Borges JB, Lubillo S, Santos A, Araujo JB, Amato MB, Suarez-Sipmann F; Open Lung Approach Network. Open Lung Approach for the Acute Respiratory Distress Syndrome: A Pilot, Randomized Controlled Trial. Crit Care Med. 2016 Jan;44(1):32-42. doi: 10.1097/CCM.0000000000001383. PMID 26672923